CLINICAL TRIAL: NCT06955754
Title: Relative Bioavailability of Three Different Oral Formulations of BI 764198 Including the Investigation of Food Effect on the Tablet Formulation in Healthy Male and Female Subjects (an Open-label, Randomised, Four-way Crossover Trial)
Brief Title: A Study in Healthy People to Test How 3 Different Formulations of BI 764198 Are Taken up in the Body and How This is Influenced by Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1434-0006; 2024-519615-34-00 (EU CTIS Number); U1111-1316-1438 (Registry Identifier: WHO - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment sequence A (Experimental): T1 - test treatment 1: BI 764198 formulation 2 administered to subjects in fasting state T2 - test treatment 2: BI 764198 formulation 2 administered to subjects after a high-fat, high-calorie breakfast T3 - test treatment 3: BI 764198 formulation 3 administered to subjects in fasting state R - reference treatment: BI 764198 formulation 1 administered to subjects in fasted state
  Interventions: Drug: BI 764198, formulation 1; Drug: BI 764198, formulation 2; Drug: BI 764198, formulation 3
- Treatment sequence B (Experimental): T2 - test treatment 2: BI 764198 formulation 2 administered to subjects after a high-fat, high-calorie breakfast T1 - test treatment 1: BI 764198 formulation 2 administered to subjects in fasting state R - reference treatment: BI 764198 formulation 1 administered to subjects in fasted state T3 - test treatment 3: BI 764198 formulation 3 administered to subjects in fasting state
  Interventions: Drug: BI 764198, formulation 1; Drug: BI 764198, formulation 2; Drug: BI 764198, formulation 3
- Treatment sequence C (Experimental): T3 - test treatment 3: BI 764198 formulation 3 administered to subjects in fasting state R - reference treatment: BI 764198 formulation 1 administered to subjects in fasted state T1 - test treatment 1: BI 764198 formulation 2 administered to subjects in fasting state T2 - test treatment 2: BI 764198 formulation 2 administered to subjects after a high-fat, high-calorie breakfast
  Interventions: Drug: BI 764198, formulation 1; Drug: BI 764198, formulation 2; Drug: BI 764198, formulation 3
- Treatment sequence D (Experimental): R - reference treatment: BI 764198 formulation 1 administered to subjects in fasted state T3 - test treatment 3: BI 764198 formulation 3 administered to subjects in fasting state T2 - test treatment 2: BI 764198 formulation 2 administered to subjects after a high-fat, high-calorie breakfast T1 - test treatment 1: BI 764198 formulation 2 administered to subjects in fasting state
  Interventions: Drug: BI 764198, formulation 1; Drug: BI 764198, formulation 2; Drug: BI 764198, formulation 3

INTERVENTIONS:
Drug: BI 764198, formulation 1 — BI 764198, formulation 1
Drug: BI 764198, formulation 2 — BI 764198, formulation 2
Drug: BI 764198, formulation 3 — BI 764198, formulation 3

SUMMARY:
This trial aims to investigate the relative bioavailability of three different oral formulations of BI 764198 and how this is influenced by food.

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m² (inclusive)
* Signed and dated written informed consent in accordance with the International Council for Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial Further inclusion criteria apply.

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 4 days
Maximum measured concentration of the analyte in plasma (Cmax) | up to 4 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 4 days
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point, dose normalized (AUC0-tz, norm) | up to 4 days
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity, dose normalized (AUC0-∞, norm) | up to 4 days
Maximum measured concentration of the analyte in plasma, dose normalised (Cmax, norm) | up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach/Riss, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com